CLINICAL TRIAL: NCT05910749
Title: Brain and Behavioral Regulation Processes in a Population With Substance Use Disorder
Brief Title: Substance Use Disorder, Brain and Behavioral Regulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not carried out because it was not approved by NIH.
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PuertoRico
Record Dates: First submitted 2023-03-27; First posted 2023-06-20 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Pre-experimental repeated measured design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- QEEG-guided sLoreta Neurofeedback (Experimental): Brainmaster Discovery 24 EEG amplifier and BrainAvatar software will be used to conduct the neurofeedback sessions
  Interventions: Device: QEEG-Guided sLoreta Neurofeedback Training

INTERVENTIONS:
Device: QEEG-Guided sLoreta Neurofeedback Training — The team will produce a neurofeedback (NFB) protocol based on QEEG sLORETA Brodmann Voxel evaluation of brain deviated/dysregulated areas. Subsequent 12 to15 sessions of individualized NFB protocol will be conducted using BrainAvatar software to normalize these regions. The NFB session will display the cortical surface and subsurface networks being trained in a live fashion. Patients will be seated on a comfortable chair in a dimly lit room and, wearing a 19-channel EEG-cap connected to an EEG amplifier, they will receive auditory and visual feedback when they meet Brodmann Voxels Z-Scores inside of +/-1.5 standard deviations (SD) on each electrode training site. Thresholds for the feedback will be first set a +/-2 SD and brought down to +/-1.5 SD throughout the sessions (subject performance dependent). Patients are encouraged to relax, hear the sounds, and watch a feedback game.

SUMMARY:
The proposed project seeks to explore the effects of a neuroregulation paradigm named Z-Score Quantitative Electroencephalogram (QEEG) guided sLORETA neurofeedback (ZQLN) on optimizing brain electrophysiological activity and behavioral performance in a substance use disorder (SUD) population whose primary drug of use is cocaine.

DETAILED DESCRIPTION:
Aim 1. Measure the effects of ZQLN training on brain electrophysiological activation changes in SUD patients. QEEG and Event-Related Potentials procedures, recorded with a 19-channel digital EEG, will be conducted before and after 12-15 sessions of ZQLN to examine changes on dysregulated brain sites by inspection of the brain maps deviating brain areas sLORETA Brodmann Areas Voxels Z-Scores inside and outside the target window of -/+2 standard deviations. Observation of P300 component latencies and amplitudes will be measured during a Drug-cue GoNoGo paradigm.

Aim 2. Measure the effects of ZQLN training on behavioral performance changes in SUD patients. In the same participants of Aim 1, Pre and Post behavioral performance (before and after 12-15 sessions of ZQLN) includes the assessment of attention and executive function, episodic memory, working memory language, and processing speed as measured by the NIH Toolbox Cognitive Domains battery scales. Other behavioral variables include reaction times, omission, and commission errors in the Drug-cue GoNoGo task.

ELIGIBILITY:
Inclusion criteria

* Age limit: 21 to 51
* Cocaine as a primary drug of selection
* Be stable (such as not having reading or movement problems preventing them from using a computer keyboard or iPad).
* Have completed the first stage of treatment in the program (this first phase consists of the stabilization and detoxification period of the program participants)

Exclusion criteria

* History of brain injury.
* Previous experience with neurofeedback training.
* Being unavailable to complete assessments.

Ages: 21 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
sLORETA Brodmann Areas Voxels Z-Scores | 2 months
  An increase of the percent of sLORETA Brodmann Areas Voxels Z-Scores inside the target window of -/+2 standard deviations after a series of ZQLN sessions is expected.
Event-Related Potentials P300 latencies | 2 months
  Brain response P300 component average latencies (measured in milliseconds) Drug-cue GoNoGo task.
Event-Related Potentials P300 amplitudes Drug-cue Go | 2 months
  Brain response P300 component average amplitudes (measured in microvolts) during Drug-cue GoNoGo. task.

SECONDARY OUTCOMES:
Attentional Executive Functioning NIH Toolbox Task | 2 months
  Flanker Inhibitory Control and Attention Task. The allocation of one's limited capacities to deal with abundance of environmental stimulation (duration 3 minutes)
Episodic Memory NIH Toolbox Task | 2 months
  Picture Sequence Memory Task. Cognitive processes involved in the acquisition, storage and retrieval of new information. (7 minutes duration)
Working Memory NIH Toolbox Task | 2 months
  List Sorting Working Memory Task. The ability to store information until the amount of information to be stored exceeds one's capacity to hold that information. (7 minutes duration)
Executive Function NIH Toolbox Task | 2 months
  Dimensional Change Card Sort Task. The capacity to plan, organize, and monitor the executive of behaviors that are strategically directed in a goal-oriented manner. (4 minutes duration)
Processing Speed NIH Toolbox Task | 2 months
  Pattern Comparison Processing Speed Test. Assesses the amount of information that can be processed within a certain unit of time. Items are simple so as to purely measure processing speed. (3 minute duration)
Drug-cue Go Task Reaction Times | 2 months
  Average Reaction times (measured in milliseconds) to the Go stimulus. In the first block of the task the Go stimulus will be a neutral category (animal or household) and in the second block the Go stimulus will be the drug-related picture.
Drug-cue Go Task Omission Errors | 2 months
  Average frequency of omission errors (not responding to the Go stimulus). In the first block of the task the Go stimulus will be a neutral category (animal or household) and in the second block the Go stimulus will be the drug-related picture.
Drug-cue NoGo Task Commission Errors | 2 months
  Average frequency of commission errors (responding to the NoGo stimulus). In the first block of the task the Go stimulus will be a neutral category (animal or household) and in the second block the Go stimulus will be the drug-related picture.

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Castillo Reyes, PhD, Principal Investigator — University of Puerto Rico
Locations (1):
- Administración de Servicios de Salud Mental y Contra la Adicción. Centro Residencial de Mujeres y Varones, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Data and findings will be published in peer-review health sciences journals and presented at national and international scientific conferences, especially those related to Neurotherapy, cognitive neuroscience, and biological psychiatry. Findings and insights gained from this study will be shared with government agencies, and medical institutions that provide services for neuro and psychiatric patients, both in Puerto Rico and in the U.S. General Data, without personal identifiers, will be made available to other researchers in Puerto Rico and other institutions outside the country for secondary analyses in their areas of expertise, or confirmation of the adequacy of our findings and conclusions. The research resources developed during the proposed project will be readily available for research purposes to qualified individuals within the scientific community to advance further research in this field. Findings will also be shared via newspapers, news releases, and press conferences.
Supporting Information: Study Protocol
Time Frame: Data will be available for one year after the study completion.
Access Criteria: Email to ismael.castillo@upr.edu